CLINICAL TRIAL: NCT05980481
Title: A Study of RC48-ADC Combine With Toripalimab and Chemotherapy or RC48-ADC Combine With Toripalimab and Trastuzumab as First-line Treatment in Local Advanced or Metastatic Gastric Cancer With the HER2 Expression or Non-expression
Brief Title: A Study of RC48-ADC Combination Therapies as First-line Treatment in Advanced Metastatic Gastric Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C027
Record Dates: First submitted 2023-07-01; First posted 2023-08-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — disitamab vedotin; Trastuzumab; toripalimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- RC48-ADC+Toripalimab+CAPOX (HER2-high expression) (Experimental): Participants with HER2-high expression(IHC2+FISH+ or IHC3+) will receive of RC48-ADC every 2 weeks (Q2W), Toripalimab every 2 weeks (Q2W) and CAPOX every 3 weeks (Q3W) , as one treatment period until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC（2.5mg/kg）; Drug: Toripalimab; Drug: Oxaliplatin（130mg/m2 ）; Drug: Capecitabine（1000mg/m2）
- RC48-ADC+Toripalimab+Trastuzumab (HER2-high expression) (Experimental): Participants with HER2-high expression(IHC2+FISH+ or IHC3+) will receive of RC48-ADC every 2 weeks (Q2W), Toripalimab every 2 weeks (Q2W) and Trastuzumab every 3 weeks (Q3W) , as one treatment period until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC（2.5mg/kg）; Drug: Trastuzumab; Drug: Toripalimab
- RC48-ADC+Toripalimab+CAPOX (HER2-intermediate/low expression) (Experimental): Participants with HER2-intermediate/low expression (IHC 2+/FISH- or IHC 1+) will receive of RC48-ADC every 2 weeks (Q2W), Toripalimab every 2 weeks (Q2W) and CAPOX every 3 weeks (Q3W) , as one treatment period until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC（2.5mg/kg）; Drug: Toripalimab; Drug: Oxaliplatin（130mg/m2 ）; Drug: Capecitabine（1000mg/m2）; Drug: RC48-ADC（2.0mg/kg）; Drug: Capecitabine（750mg/m2）; Drug: Oxaliplatin（100mg/m2 ）
- Toripalimab+Trastuzumab+CAPOX (HER2-high expression) (Active Comparator): Participants with HER2-high expression (IHC2+FISH+ or IHC3+) will receive of Toripalimab every 2 weeks (Q2W) , Trastuzumab every 3 weeks (Q3W) and CAPOX every 3 weeks (Q3W) , as one treatment period until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Trastuzumab; Drug: Toripalimab; Drug: Oxaliplatin（130mg/m2 ）; Drug: Capecitabine（1000mg/m2）
- Toripalimab+CAPOX (HER2- intermediate/low expression) (Active Comparator): Participants with HER2- intermediate/low expression (IHC 2+/FISH- or IHC 1+) will receive of Toripalimab every 2 weeks (Q2W) and CAPOX every 3 weeks (Q3W) , as one treatment period until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Toripalimab; Drug: Oxaliplatin（130mg/m2 ）; Drug: Capecitabine（1000mg/m2）
- RC48-ADC + Toripalimab + Trastuzumab + Capecitabine (HER2-high expression) (Experimental): Participants with HER2-high expression(IHC2+FISH+ or IHC3+) will receive of RC48-ADC every 2 weeks (Q2W), Toripalimab every 2 weeks (Q2W) , Trastuzumab every 3 weeks (Q3W) and Capecitabine every 3 weeks (Q3W), as one treatment period until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC（2.5mg/kg）; Drug: Trastuzumab; Drug: Toripalimab; Drug: Capecitabine（1000mg/m2）
- RC48-ADC+Toripalimab+CAPOX (HER2-negative) (Experimental): Participants with HER2-negative (IHC0) will receive of RC48-ADC every 2 weeks (Q2W), Toripalimab every 2 weeks (Q2W) and CAPOX every 3 weeks (Q3W) , as one treatment period until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC（2.5mg/kg）; Drug: Toripalimab; Drug: RC48-ADC（2.0mg/kg）; Drug: Capecitabine（750mg/m2）; Drug: Oxaliplatin（100mg/m2 ）
- Toripalimab+CAPOX (HER2- negative) (Active Comparator): Participants with HER2- negative (IHC 0) will receive of Toripalimab every 2 weeks (Q2W) and CAPOX every 3 weeks (Q3W) , as one treatment period until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Toripalimab; Drug: Oxaliplatin（130mg/m2 ）; Drug: Capecitabine（1000mg/m2）

INTERVENTIONS:
Drug: RC48-ADC（2.5mg/kg） — 2.5 mg/kg intravenous infusion every 2 weeks
  Other Names: Disitamab Vedotin
  Arms: RC48-ADC + Toripalimab + Trastuzumab + Capecitabine (HER2-high expression); RC48-ADC+Toripalimab+CAPOX (HER2-high expression); RC48-ADC+Toripalimab+CAPOX (HER2-intermediate/low expression); RC48-ADC+Toripalimab+CAPOX (HER2-negative); RC48-ADC+Toripalimab+Trastuzumab (HER2-high expression)
Drug: Trastuzumab — First load dose is 8.0mg , then 6.0 mg/kg intravenous infusion every 3 weeks
  Other Names: Trastuzumab Injection
  Arms: RC48-ADC + Toripalimab + Trastuzumab + Capecitabine (HER2-high expression); RC48-ADC+Toripalimab+Trastuzumab (HER2-high expression); Toripalimab+Trastuzumab+CAPOX (HER2-high expression)
Drug: Toripalimab — 3.0 mg/kg intravenous infusion every 2 weeks
  Other Names: JS001
Drug: Oxaliplatin（130mg/m2 ） — 130mg/m2 intravenous infusion Q3W
  Other Names: Oxaliplatin injection
  Arms: RC48-ADC+Toripalimab+CAPOX (HER2-high expression); RC48-ADC+Toripalimab+CAPOX (HER2-intermediate/low expression); Toripalimab+CAPOX (HER2- intermediate/low expression); Toripalimab+CAPOX (HER2- negative); Toripalimab+Trastuzumab+CAPOX (HER2-high expression)
Drug: Capecitabine（1000mg/m2） — 1000mg/m2 per os Q3W
  Other Names: Capecitabine Tablets
  Arms: RC48-ADC + Toripalimab + Trastuzumab + Capecitabine (HER2-high expression); RC48-ADC+Toripalimab+CAPOX (HER2-high expression); RC48-ADC+Toripalimab+CAPOX (HER2-intermediate/low expression); Toripalimab+CAPOX (HER2- intermediate/low expression); Toripalimab+CAPOX (HER2- negative); Toripalimab+Trastuzumab+CAPOX (HER2-high expression)
Drug: RC48-ADC（2.0mg/kg） — 2.0 mg/kg intravenous infusion every 2 weeks
  Other Names: Disitamab Vedotin
  Arms: RC48-ADC+Toripalimab+CAPOX (HER2-intermediate/low expression); RC48-ADC+Toripalimab+CAPOX (HER2-negative)
Drug: Capecitabine（750mg/m2） — 750mg/m2 per os Q3W
  Other Names: Capecitabine Tablets
  Arms: RC48-ADC+Toripalimab+CAPOX (HER2-intermediate/low expression); RC48-ADC+Toripalimab+CAPOX (HER2-negative)
Drug: Oxaliplatin（100mg/m2 ） — 100mg/m2 intravenous infusion Q3W
  Other Names: Oxaliplatin injection（100mg/m2 ）
  Arms: RC48-ADC+Toripalimab+CAPOX (HER2-intermediate/low expression); RC48-ADC+Toripalimab+CAPOX (HER2-negative)

SUMMARY:
This is a Phase II/III, randomized, multicenter, open-label clinical trial designed to evaluate safety and efficacy of RC48-ADC combine with Toripalimab and chemotherapy or RC48-ADC combine with Toripalimab and Trastuzumab as first-line treatment in human epidermal growth factor receptor 2 (HER2)-expression or non-expression participants with locally advanced or metastatic gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Age:18-75 years（including 18 and 75）.
* Predicted survival ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function.
* All subjects must have inoperable, advanced or metastatic gastric or or gastroesophageal adenocarcinoma.
* Subject must be previously untreated with systemic treatment; Subject that received neoadjuvant chemotherapy with recurrence >6 months from completion of therapy are permitted;
* HER2-expressing status determined by laboratory to be IHC 1+, 2+ or 3+ or IHC0.

Exclusion Criteria:

* Active central nervous system (CNS) metastases.
* Known active hepatitis B, active hepatitis C, or human immunodeficiency virus (HIV) infection.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, thyroid cancer ,etal.
* Known hypersensitivity to antibody-drug conjugate(ADC) or PD-(L)1 or any of its components.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years
  The objective response rate will be mainly analyzed by according to the RECIST 1.1 standard tumor evaluation by the investigator will be performed).

SECONDARY OUTCOMES:
Safety(adverse event) | Up to approximately 2 years
  to evaluate safety including adverse event rate and adverse event grade.
Progression-free survival (PFS), evaluated by the investigator | Up to approximately 2 years
  Progression-free survival (PFS) refers to the time from the date of randomization to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard.
Overall survival (OS) | Up to approximately 2 years
  Overall survival (OS) refers to the time from the date of randomization to the date of death of the subject.
Duration of response (DOR) | Up to approximately 2 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death
Disease Control Rate(DCR) | Up to approximately 2 years
  DCR is the proportion of subjects with optimal overall response to achieve objective remission or stable disease over the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Na Su, PhD, Study Director — RemeGen Co., Ltd.
Locations (1):
- Beijing Cancer Hospital, Beijing, China